CLINICAL TRIAL: NCT03612635
Title: Impact on Patient Outcome and Healthcare Utilization of Cardiac ImplaNTable Electronic Devices Complications
Brief Title: Impact on Patient Outcome of Cardiac Implantable Electronic Device Complications
Acronym: POINTED
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Cardinale G. Panico (Other)
Responsible Party: Sponsor
Other Study IDs: POINTED
Record Dates: First submitted 2018-07-19; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Cardiac Implantable Electronic Device Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Implantation of a cardiac implantable electronic device — All patients enrolled in the registry underwent cardiac implantable electronic device implantation

SUMMARY:
The purpose of this registry is to evaluate the impact on patient outcome and on healthcare utilization of cardiac implantation electronic device complications during a long-term follow-up.

DETAILED DESCRIPTION:
Multicentric, observational, prospective registry enrolling consecutive patients underwent pacemaker or defibrillator implantation, aimed to evaluate the impact of cardiac implantable device complications requiring surgical revision on healthcare utilization (number and length of hospitalizations), and on patient outcome (all-cause mortality and cardiac mortality), during a long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent cardiac implantable electronic device implantation according to current guidelines during the enrollment period.

Exclusion Criteria:

* patients already carriers of a cardiac implantable electronic device underwent replacement or upgrading of device.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with indication to receive a cardiac implantable electronic device (pacemaker or defibrillator).
Sampling Method: Non-Probability Sample
Enrollment: 2811 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
All-cause Death (dead/alive status assessment during follow-up) | An average of 48 months
  Evaluation of all-cause mortality during follow-up

SECONDARY OUTCOMES:
Occurrence of hospitalizations related to cardiac implantable electronic device complications | An average of 48 months
  Evaluation of hospitalizations related to cardiac implantable electronic device complications

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - "Card. G. Panico" Hospital, Tricase, Lecce
  - Federico Guerra, Ancona
  - Policlinico S.Orsola-Malpighi, Bologna
  - Mattia Laffi, Genova
  - Monaldi Hospital, Napoli
  - AOU "Maggiore della Carità", Novara

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Palmisano P, Sergi C, Panico V, Chiarillo MV, Chiuri MD, Martella ML, Stefanelli G, Martella D, Mauro R, Ponzetta MA, Parlavecchio A, Accogli M, Coluccia G. Impact on nurse workload and patient satisfaction of atrioventricular junction ablation performed simultaneously with conduction system pacing using a superior approach from the pocket compared with the conventional femoral approach. Eur J Cardiovasc Nurs. 2024 Oct 21;23(7):746-755. doi: 10.1093/eurjcn/zvae043. PMID 38552177